CLINICAL TRIAL: NCT03306355
Title: Clinical Study to Compare Clinical Outcomes of IOLs FineVision POD F GF (Hydrophobic) and FineVision POD F (Hydrophilic) After Bilateral Implantation in Asian Eyes
Brief Title: Comparison of Clinical Outcomes on Trifocal IOLs FineVision POD F GF and FineVision POD F in Asian Eyes
Acronym: PHY1706
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHY 1706
Record Dates: First submitted 2017-09-28; First posted 2017-10-11 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular Lens; trifocal; hydrophobic; hydrophilic
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL implantation experimental (Experimental): hydrophobic, trifocal intraocular lens POD F GF
  Interventions: Device: IOL implantation experimental
- IOL implantation active comparator (Active Comparator): hydrophilic, trifocal intraocular lens POD F
  Interventions: Device: IOL implantation active comparator

INTERVENTIONS:
Device: IOL implantation experimental — Implantation of trifocal IOL POD F GF consisting of hydrophobic material
  Arms: IOL implantation experimental
Device: IOL implantation active comparator — Implantation of trifocal IOL POD F consisting of hydrophilic material
  Arms: IOL implantation active comparator

SUMMARY:
Prospective, randomised, controlled, single-surgeon, single-center clinical study to compare the clinical outcomes of two trifocal IOLs with different material (hydrophobic and hydrophilic) from the same manufacturer. Implantation of the IOLs is bilaterally.

DETAILED DESCRIPTION:
This is a prospective, randomised, controlled, single-surgeon, single-center clinical study whereby patients undergoing routine cataract surgery will have bilateral implantation of trifocal intraocular lenses. The patients will either be implanted with the hydrophobic IOL FineVision POD F GF or the hydrophilic IOL FineVision POD F (both lenses: (PhysIOL, Liège, Belgium).

The devices under investigation (FineVision POD F GF and POD F) are trifocal glistening-free acrylic intraocular lenses (IOLs) manufactured by the sponsor of this study PhysIOL sa/nv. The main difference between the lenses is the material (hydrophobic and hydrophilic). The IOLs will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

Subjects participating in the trial will attend a total of 12 study visits (1 preoperative, 2 operative and 9 postoperative) over a period of 36 months. Subjects would have the option for unscheduled visits if required medically.

Primary endpoint data will be collected at the 3 months follow up visit and secondary endpoint data will be collected at the 3, 12, 24 and 36 months follow up visits. Data analyses will be done after the last patient finished the final examination to support the study publication plan.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity
* Spontaneously emitting the desire for spectacle independence after surgery and with realistic expectation.
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Unrealistic expectation
* Age of patient <45 years
* Irregular astigmatism
* Regular corneal astigmatism >0.75 dioptres by an automatic keratometer or biometer or >1.0 dioptres if the steep axis of cylinder is between 90° and 120°
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* Age-related Macular Degeneration (AMD) suspicious eyes (determined by OCT)
* Complicated surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions. | 3 months postoperative
  No statistically significant difference between the two study groups on monocular UDVA at 3 months follow up visit. A significance level of 0.05 or lower (p < 0.05) will be considered statistically significant. UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014

SECONDARY OUTCOMES:
Manifested refraction | Pre-OP, 1 week postoperative, 1 month postoperative, 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2014. This data will also be used to calculate the manifested refractive spherical equivalent (MRSE)
Uncorrected Distance Visual Acuity (UDVA) - monocular | 1 day postoperative, 1 week postoperative, 1 month postoperative, 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly.
Uncorrected Distance Visual Acuity (UDVA) - binocular | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done binocularly.
Corrected Distance Visual Acuity (CDVA) - monocular | Pre-OP, 1 week postoperative, 1 month postoperative, 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done monocularly.
Corrected Distance Visual Acuity (CDVA) - binocular | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done binocularly.
Distance Corrected Intermediate Visual Acuity at 70cm (DCIVA) - monocular | 1 week postoperative, 1 month postoperative, 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  DCIVA is measured with ETDRS charts placed in 70cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly.
Distance Corrected Intermediate Visual Acuity at 70cm (DCIVA) - binocular | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  DCIVA is measured with ETDRS charts placed in 70cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done binocularly.
Uncorrected Intermediate Visual Acuity at 70cm (UIVA) - monocular | 1 week postoperative, 1 month postoperative, 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  UIVA is measured with ETDRS charts placed in 70cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly.
Uncorrected Intermediate Visual Acuity at 70cm (UIVA) - binocular | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  UIVA is measured with ETDRS charts placed in 70cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done binocularly.
Distance Corrected Near Visual Acuity at 35cm (DCNVA) - monocular | 1 week postoperative, 1 month postoperative, 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly.
Distance Corrected Near Visual Acuity at 35cm (DCNVA) - binocular | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done binocularly.
Uncorrected Near Visual Acuity at 35cm (UNVA) | 1 week postoperative, 1 month postoperative, 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  UNVA is measured with ETDRS charts placed in 35cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly.
Uncorrected Near Visual Acuity at 35cm (UNVA) | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  UNVA is measured with ETDRS charts placed in 35cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done binocularly.
Contrast Sensitivity | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  Contrast Sensitivity under photopic and mesopic light conditions
Aberrometry | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  Aberrometry outcomes are measured with a standard aberrometer. The following values will be evaluated in this study: Spherical aberrations, high order aberrations, lens tilt.
AcuTarget diagnostic device | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  Measurement of Ocular Scatter Index (OSI) score to evaluate and compare the scattering of the implanted lenses.
Visual Functioning Questionnaire - 25 (VFQ-25) | 3 months postoperative, 12 months postoperative.
  Outcomes measures of a questionnaire to address the general patient satisfaction and possible side effects of the treatment. For this study, the validated and verified Visual Functioning Questionnaire - 25 (VFQ-25) will be used. The maximum score for each questionaire is 100.
Defocus Curve | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -5.0 D to +1.5 D. This examination is performed monocularly and binocularly.
Slitlamp examination - Corneal Status | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Slitlamp examination - Fundus | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slitlamp examination - Signs of inflammation | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Signs of inflammation
Slitlamp examination - Pupillary block | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Pupillary block
Slitlamp examination - Retinal detachment | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Retinal detachment
Slitlamp examination - Status of anterior and posterior capsule | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Status of anterior and posterior capsule
Slitlamp examination - IOL decentration | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL decentration
Slitlamp examination - IOL tilt | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL tilt
Slitlamp examination - IOL discoloration | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL discoloration
Slitlamp examination - IOL opacity | 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL opacity

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | Pre-OP, 1 day postoperative, 1 week postoperative, 1 month postoperative, 3 months postoperative, 12 months postoperative, 24 months postoperative, 36 months postoperative.
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations
Keratometry | Pre-OP
  Keratometric measurements are performed to calculate the required IOL power
Biometry | Pre-OP
  Biometry measurements are performed to calculate the required IOL power

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edward Ang, MD, Principal Investigator — Asian Eye Institute
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: No